CLINICAL TRIAL: NCT05762458
Title: Efficacy and Safety of Ammoxetine Hydrochloride Enteric-coated Tablets in Subjects With Depression: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Phase Ⅱ Study
Brief Title: The Study of Ammoxetine Hydrochloride Enteric-coated Tablets in Subjects With Depression
Acronym: Ammoxetine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HA1406-005
Record Dates: First submitted 2023-01-28; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-01

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: MDD
MeSH Terms: conditions — Depressive Disorder, Major | interventions — ammoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ammoxetine group-cohort 1 (Experimental): The eligible subjects will receive Ammoxetine hydrochloride enteric-coated tablets plus placebo.
  Interventions: Drug: Ammoxetine; Drug: Placebo
- Ammoxetine group-cohort 2 (Experimental): The eligible subjects will receive Ammoxetine hydrochloride enteric-coated tablets plus placebo.
  Interventions: Drug: Ammoxetine; Drug: Placebo
- Placebo group (Placebo Comparator): The eligible subjects will receive placebo to Ammoxetine.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ammoxetine — Ammoxetine hydrochloride enteric-coated tablets
  Arms: Ammoxetine group-cohort 1; Ammoxetine group-cohort 2
Drug: Placebo — placebo to Ammoxetine.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Ammoxetine hydrochloride enteric-coated tablets in subjects with depression.

DETAILED DESCRIPTION:
In this study, a randomized, double-blind, placebo-controlled multicenter study will be conducted to evaluate the efficacy and safety of different doses of Ammoxetine hydrochloride enteric coated tablets in the treatment of depression.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 and 65 years (inclusive), no gender limitation;
2. Subject has recurrent Major Depressive Disorder (MDD) as the primary diagnosis according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5, 5th Edition), single episode or recurrent episodes (DSM-IV-TR criteria, classification code 296.2/296.3), without psychotic symptoms;
3. Subjects with a Montgomery-Asberg Depression Rating Scale (MADRS) score ≥ 26 at screening and baseline;
4. Subjects with Clinical Global Impression Scale Disease Severity CGI-S severity score ≥ 4 at screening and baseline;
5. A score of ≥2 on the first item (depressed mood) of the HAMD-17 scale at the screening and baseline;
6. Male or female with fertility must agree to use effective contraceptive method during the study and within 1 month after the end of the trial;
7. Be able to read and understand the content of the informed consent and voluntarily sign the informed consent.

Exclusion Criteria:

1. Subjects with ≥ 25% reduction in MADRS score in the baseline period compared to the screening period;
2. Subjects meet DSM-5 diagnostic criteria for other mental disorders (schizophrenia spectrum and other psychiatric disorders, bipolar and related disorders, anxiety disorders, obsessive-compulsive and related disorders, somatic symptoms and related disorders, etc.);
3. Subjects are diagnosed as DSM-5 drug use disorder;
4. Refractory depression (subjects who had previously used two different mechanisms of antidepressants and failed after receiving adequate treatment (at least 8 weeks);
5. Organic mental disorders, such as depression caused by hypothyroidism;
6. Depression caused by psychoactive substances or non-addictive substances;
7. Subjects with other diseases or other types of mental disorders with depressive symptoms;
8. Subjects assessed by the Columbia Suicide Severity Rating Scale (C-SSRS) and those judged by the investigator to be at risk for suicide, or to have engaged in suicidal behavior within 6 months prior to screening;
9. Allergic constitution (e.g. allergic to two or more drugs or to serotonin norepinephrine reuptake inhibitors (SNRIs));
10. Previous history of malignant tumor;
11. Previous history of elevated intraocular pressure or narrow angle glaucoma;
12. Subjects suffered from other serious physical diseases, such as uncontrolled hypertension or unstable cardiovascular disease, serious liver disease, kidney disease, blood disease, endocrine disease, neurological disease, etc;
13. Subjects with diseases that interfere with the absorption of oral medications, such as active bowel disease, partial or complete intestinal obstruction, chronic diarrhea, etc;
14. Subjects who have used drugs or foods that alter the activity of liver enzymes (CYP2C19 and CYP3A4) such as dexamethasone, rifampicin, omeprazole, etc., within 4 weeks prior to randomization;
15. 12-lead ECG system showed degree Ⅱ or Ш atrioventricular block, long QT syndrome or QTc > 450 ms (male) / 460 ms (female) at screening;
16. Subjects discontinued use of a combination of drugs that prolong the QT interval prior to randomization, or drugs that can cause prolongation of the QT and may induce TdP for less than 5 half-lives of the drugs;
17. In screening period, subjects with ALT or AST 2 times higher than the upper limit of laboratory normal value; and abnormalities in 2 or more of the 5 indicators of thyroid function (TSH, FT3, FT4, TT3 or TT4 0.9 times below the lower limit of normal value or 1.1 times above the upper limit of normal value);
18. Subjects have used monoamine oxidase inhibitors within 2 weeks before randomization;
19. Subjects discontinuing antipsychotics, antidepressants or mood stabilizers for less than 5 half-lives of the drug before randomization;
20. Subjects who are using long half-life drugs (such as fluoxetine, long-acting antipsychotics, etc.);
21. Subjects who have received electroconvulsive therapy (ECT), systematic psychotherapy (interpersonal relationship therapy, dynamic therapy, cognitive behavior therapy, etc.), transcranial magnetic stimulation (TMS), vagus nerve stimulation (VNS), phototherapy, etc. within 3 months before screening, or subjects who, in the judgment of the investigator, are currently in need of such treatment;
22. Female subjects who are breastfeeding or have a positive pregnancy test during the screening period or during the study;
23. Alcohol or drug dependence within 3 months before screening;
24. Subjects who have participated in other clinical trials within 3 months before screening and are taking the test drug;
25. Subjects who, in the opinion of the investigator, have any other condition that makes them unsuitable for participation in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-02-28 (Estimated); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Montgomery Asperger Depression Scale (MADRS) score at the end of treatment (week 8) | Baseline and week 8
  The MADRS is a clinician-rated scale to assess depressive symptomatology during the preceding week. Participants are rated on 10 items (feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and lack of interest) each on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). The total score ranges from 0 to 60 with a higher score indicating more depression. A negative change score indicates improvement.

SECONDARY OUTCOMES:
Change from baseline in Hamilton Depression Scale (HAMD-17) at week 1, 2, 4, 6, 8 | Baseline, week 1, 2, 4 ,6 and 8
Change from baseline in Hamilton Anxiety Inventory (HAMA) scores at week 1, 2, 4, 6, 8 | Baseline, week 1, 2, 4 ,6 and 8
Change from baseline in CGI-S score at week 1, 2, 4, 6, 8 | Baseline, week 1, 2, 4, 6 and 8
Change from baseline in MADRS score at week 1, 2, 4, 6 | baseline, week 1, 2 and 4, 6
CGI-I scores at the end of 8 weeks of treatment at week 1, 2, 4, 6, 8 | Baseline, week 1, 2, 4, 6 and 8
The efficiency and remission of the MADRS score | Baseline, Baseline, week 1, 2, 4, 6 and 8
  Effectiveness is defined as ≥ 50% reduction in MADRS score relative to baseline after treatment. Remission is defined as ≤ 10 MADRS score after treatment.
Efficacy and remission of HAMD-17 scores | Baseline, week 1, 2, 4, 6 and 8
  Effectiveness is defined as ≥50% reduction in HAMD-17 score relative to baseline after treatment. Remission is defined as HAMD-17 score ≤7 after treatment.
The percentage of subjects with a MARDS score reduction ≥ 25% | Week 1 and 2
Incidence of adverse events (AE) | Throughout the study period（From baseline to week 10）

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] He S, Chen JX, Yu X, Lin H, Wang Z, Li X, Zhou Y, Liu YS, Zhang H, Wang J, An C, Liu H, Li C, Ni S, Li H. Efficacy and Safety of Ammoxetine in Major Depressive Disorder: A Randomized Clinical Trial. JAMA Netw Open. 2025 Sep 2;8(9):e2532650. doi: 10.1001/jamanetworkopen.2025.32650. PMID 40982284